CLINICAL TRIAL: NCT01127698
Title: Swedish Mammography Cohort
Acronym: SMC
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Harvard School of Public Health (HSPH) (Other)
Responsible Party: Principal Investigator, Alicja Wolk, Professor, Karolinska Institutet
Other Study IDs: 1706/2010-631-1
Record Dates: First submitted 2010-05-20; First posted 2010-05-21 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-02

CONDITIONS: Cancers; Cardiovascular Diseases; Cataract; Gastrointestinal Diseases; Osteoporosis; Fractures
MeSH Terms: conditions — Neoplasms; Cardiovascular Diseases; Cataract; Gastrointestinal Diseases; Osteoporosis; Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva Blood
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The Swedish Mammography Cohort began in 1987-1990, when 66,651 women living in two counties in central Sweden completed a mailed questionnaire that included items about their diet, parity, age at first child's birth, history of breast cancer in family, weight, height, and education. Follow-up questionnaires have been sent out in 1997 and in 2008-09.

DETAILED DESCRIPTION:
From 1987 to 1990 a population-based mammography screening program was introduced in two counties in central Sweden. In Västmanland County all women born between 1917 and 1948 received a mailed invitation to be screened by mammography between March 1987 and March 1989 (n=41,786) together with a 6-page questionnaire; 31,735 women (76%) returned the completed questionnaires. In Uppsala County all women born between 1914 and 1948 were invited to the screening and received the same questionnaire between January 1988 and December 1990 (n=48517); 34916 women (72%) returned the completed questionnaires. Hence, questionnaires completed before undergoing mammography were obtained from 66,651 women (74%) in the source population. These questionnaires included items about diet, parity, age at first child's birth, history of breast cancer in family, weight, height, and education.

In 1997 a second questionnaire was sent to all cohort members who were still living in the study area. The questionnaire updated information about diet and was extended to include information on physical activity, medical history, age at menarche, history of oral contraceptive use, age at menopause, postmenopausal hormone use and lifestyle factors such as cigarette smoking history and use of dietary supplements. Majority of questions in the questionnaires have been validated.

During 2008-09, the exposure information was updated and extended by sending out two new questionnaires - one questionnaire on health including several signs of symptoms, sleeping, social relations etc (2008) and one on diet, dietary supplement use, and lifestyle factors (2009).

Incident cases of cancer are ascertained by record linkages of the study population with the National Swedish Cancer Register and the Regional Cancer Registers. Cardiovascular and other diseases as well as surgeries and causes of death are identified by linkage to the National Inpatient and other registries at the Swedish Board of Health and Welfare. Ascertainment of cancer cases and other diseases is almost 100% complete. Dates of deaths are ascertained through the Swedish Death Register (100% complete), and information on date of moving out of the study area is obtained by linkage with the Swedish Population Register.

ELIGIBILITY:
Inclusion Criteria:

* All women born between 1914 and 1948, living in central Sweden

Exclusion Criteria:

* None

Ages: 40 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women born between 1914 and 1948, living in central Sweden (Uppsala and Västmanlands counties)
Sampling Method: Non-Probability Sample
Enrollment: 61433 (Estimated)
Dates: Start 1987-03; Primary Completion 1990-12 (Actual)

PRIMARY OUTCOMES:
Breast cancer | 1987-2010
Colorectal cancer | 1987-2010
Endometrial Cancer | 1987-2010
Ovarian cancer | 1987-2010
Pancreatic cancer | 1987-2010
Stomach cancer | 1987-2010
Kidney cancer | 1987-2010
Bladder cancer | 1987-2010
Cardiovascular diseases | 1987-2010
Mortality | 1987-2010
Cataract | 1987-2010
Fractures, hip fractures | 1987-2014

REFERENCES:
- [Derived] Larsson SC, Drca N, Bjorck M, Back M, Wolk A. Nut consumption and incidence of seven cardiovascular diseases. Heart. 2018 Oct;104(19):1615-1620. doi: 10.1136/heartjnl-2017-312819. Epub 2018 Apr 16. PMID 29661934
- [Derived] Larsson SC, Wallin A, Hakansson N, Stackelberg O, Back M, Wolk A. Type 1 and type 2 diabetes mellitus and incidence of seven cardiovascular diseases. Int J Cardiol. 2018 Jul 1;262:66-70. doi: 10.1016/j.ijcard.2018.03.099. Epub 2018 Mar 24. PMID 29605469
- [Derived] Roze JC, Ancel PY, Lepage P, Martin-Marchand L, Al Nabhani Z, Delannoy J, Picaud JC, Lapillonne A, Aires J, Durox M, Darmaun D, Neu J, Butel MJ; Nutrition EPIPAGE 2 study group; EPIFLORE Study Group. Nutritional strategies and gut microbiota composition as risk factors for necrotizing enterocolitis in very-preterm infants. Am J Clin Nutr. 2017 Sep;106(3):821-830. doi: 10.3945/ajcn.117.152967. Epub 2017 Jun 28. PMID 28659297
- [Derived] Larsson SC, Wolk A. Potato consumption and risk of cardiovascular disease: 2 prospective cohort studies. Am J Clin Nutr. 2016 Nov;104(5):1245-1252. doi: 10.3945/ajcn.116.142422. Epub 2016 Sep 28. PMID 27680993
- [Derived] Bellavia A, Stilling F, Wolk A. High red meat intake and all-cause cardiovascular and cancer mortality: is the risk modified by fruit and vegetable intake? Am J Clin Nutr. 2016 Oct;104(4):1137-1143. doi: 10.3945/ajcn.116.135335. Epub 2016 Aug 24. PMID 27557655
- [Derived] Xu H, Akesson A, Orsini N, Hakansson N, Wolk A, Carrero JJ. Modest U-Shaped Association between Dietary Acid Load and Risk of All-Cause and Cardiovascular Mortality in Adults. J Nutr. 2016 Aug;146(8):1580-5. doi: 10.3945/jn.116.231019. Epub 2016 Jul 6. PMID 27385761
- [Derived] Larsson SC, Tektonidis TG, Gigante B, Akesson A, Wolk A. Healthy Lifestyle and Risk of Heart Failure: Results From 2 Prospective Cohort Studies. Circ Heart Fail. 2016 Apr;9(4):e002855. doi: 10.1161/CIRCHEARTFAILURE.115.002855. PMID 27072861
- [Derived] Larsson SC, Wallin A, Wolk A. Dietary Approaches to Stop Hypertension Diet and Incidence of Stroke: Results From 2 Prospective Cohorts. Stroke. 2016 Apr;47(4):986-90. doi: 10.1161/STROKEAHA.116.012675. Epub 2016 Feb 11. PMID 26869384
- [Derived] Larsson SC, Hakansson N, Wolk A. Dietary cysteine and other amino acids and stroke incidence in women. Stroke. 2015 Apr;46(4):922-6. doi: 10.1161/STROKEAHA.114.008022. Epub 2015 Feb 10. PMID 25669310
- [Derived] Oskarsson V, Orsini N, Sadr-Azodi O, Wolk A. Fish consumption and risk of non-gallstone-related acute pancreatitis: a prospective cohort study. Am J Clin Nutr. 2015 Jan;101(1):72-8. doi: 10.3945/ajcn.113.076174. Epub 2014 Nov 5. PMID 25527752
- [Derived] Bellavia A, Larsson SC, Bottai M, Wolk A, Orsini N. Differences in survival associated with processed and with nonprocessed red meat consumption. Am J Clin Nutr. 2014 Sep;100(3):924-9. doi: 10.3945/ajcn.114.086249. Epub 2014 Jul 16. PMID 25030780
- [Derived] Bellavia A, Larsson SC, Bottai M, Wolk A, Orsini N. Fruit and vegetable consumption and all-cause mortality: a dose-response analysis. Am J Clin Nutr. 2013 Aug;98(2):454-9. doi: 10.3945/ajcn.112.056119. Epub 2013 Jun 26. PMID 23803880
- [Derived] Genkinger JM, Friberg E, Goldbohm RA, Wolk A. Long-term dietary heme iron and red meat intake in relation to endometrial cancer risk. Am J Clin Nutr. 2012 Oct;96(4):848-54. doi: 10.3945/ajcn.112.039537. Epub 2012 Sep 5. PMID 22952183
- [Derived] Larsson SC, Virtamo J, Wolk A. Fish consumption and risk of stroke in Swedish women. Am J Clin Nutr. 2011 Mar;93(3):487-93. doi: 10.3945/ajcn.110.002287. Epub 2010 Dec 29. PMID 21191140
- See also: Unit of Nutritional Epidemiology — http://ki.se/ki/jsp/polopoly.jsp?l=en&d=20996